CLINICAL TRIAL: NCT01073488
Title: Evaluation of an Emergency Obstetric and Neonatal Care (EmONC) Intervention Package to Reduce Adverse Pregnancy Outcomes in Low Resource Settings (The EmONC Trial)
Brief Title: Emergency Obstetric and Neonatal Care: The EmONC Trial
Acronym: EmONC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GN EmONC
Record Dates: First submitted 2010-02-21; First posted 2010-02-23 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Maternal Morbidity and Mortality; Stillbirth and Neonatal Mortality
Keywords: Pregnancy; Maternal child health; Developing countries; Stillbirth; Neonatal mortality; Maternal mortality; Community intervention; Community mobilization; Home-based Life Saving Skills
MeSH Terms: conditions — Stillbirth; Maternal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EMONC: Community mobilization, HBLSS and Facility Improvement (Experimental): The intervention group received training in community mobilization activities, Home Based Life Saving Skills (HBLSS) and facility improvement.
  Interventions: Behavioral: Community Mobilization, HBLSS and facility improvement
- Control (No Intervention): The control group did not receive an intervention, but collected outcome data through a baseline maternal/newborn birth registry.

INTERVENTIONS:
Behavioral: Community Mobilization, HBLSS and facility improvement — Mobilization of the community, with special emphasis on pregnant women and their families, to identify resources and solutions to improve maternal and neonatal mortality, home-based life savings skills (HBLSS) for community birth attendants and facility improvement activities.
  Other Names: CM
  Arms: EMONC: Community mobilization, HBLSS and Facility Improvement

SUMMARY:
The objective of this cluster randomized controlled trial is to reduce maternal and neonatal mortality by increasing access to and improving the quality of obstetric and neonatal care for pregnant women in study clusters. It is hypothesized that a 25% reduction in >28 week or >1000 gram stillbirth and 7-day neonatal mortality will be achieved in the intervention clusters by a multifaceted Emergency Obstetric Neonatal Care (EmONC) package that will be introduced by an EmONC team.

DETAILED DESCRIPTION:
Maternal death, stillbirth, early neonatal death, and obstetric fistula are among the most devastating adverse outcomes of pregnancy. Existing interventions could avert the majority of maternal and neonatal deaths; however, those women at greatest risk are least likely to have access to interventions delivered through the formal health care system. In many developing countries, most deliveries in rural areas and a significant number in urban areas are conducted at home without skilled attendance, circumstances which pose a high risk for both mothers and their neonates. The EmONC trial is designed to evaluate a comprehensive intervention encompassing community mobilization to establish and sustain mechanisms of transport and payment and to drive client-oriented emergency obstetrical and neonatal care. The intervention includes teaching recognition of prolonged labor, infection, preeclampsia and hemorrhage, and the use of appropriate stabilization methods by all community birth attendants. In addition, poor access to quality emergency obstetric and neonatal care in a sustainable manner will be addressed. To evaluate the effectiveness of this approach, a cluster-randomized trial is required to assess whether Cluster EmONC teams can work with the community and health care system to reduce adverse pregnancy outcomes in diverse settings where the majority of deliveries occur at home or at a health clinic with few or no available EmONC interventions. To accomplish the intervention, a train-the-trainer approach will be used. Master trainers will facilitate central and regional training sessions for Country trainers organized around the areas of community mobilization; birth attendant skills; and EmONC referral facility improvements. The Country trainers will then support training and related activities in the intervention clusters, predominantly focusing on these three areas. The study population includes pregnant women (and their neonates) living and delivering in the 108 study clusters. The study clusters are largely rural, geographically distinct communities, each of which have approximately 300 annual deliveries. The women will be enrolled at or after 20 weeks gestation and followed to 42 days post delivery. The total duration of the trial will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women living in and/or delivering within the study cluster
2. Consent provided

Exclusion Criteria: Eligible pregnant women who do not consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 267181 (Actual)
Dates: Start 2008-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Composite of either >28 week / >1000 gram stillbirth or 7 day neonatal mortality rate | 7 days post delivery

SECONDARY OUTCOMES:
Maternal mortality rate | 42 days post delivery
Maternal morbidity rates | 42 days post delivery
Stillbirth rate | Delivery
7-day neonatal mortality rate | 7 days post delivery
28-day neonatal mortality rate | 28 days post delivery
Rates of mothers transported to a referral hospital. | 42 days post delivery
Rates of neonates/infants transported to a referral hospital | 42 days post delivery

CONTACTS AND LOCATIONS:
Overall Officials: Robert Goldenberg, MD, Principal Investigator — Drexel University College of Medicine
Locations (7):
- University of Buenos Aires, Buenos Aires, Argentina
- IMSALUD / San Carlos University, Guatemala City, Guatemala
- India (2):
  - Jawaharlal Nehru Medical College, Belagavi
  - Indira Gandhi Government Medical College, Nagpur
- Moi University School of Medicine, Eldoret, Kenya
- The Aga Khan University, Karachi, Pakistan
- University Teaching Hospital, Lusaka, Zambia

REFERENCES:
- [Derived] Pasha O, McClure EM, Wright LL, Saleem S, Goudar SS, Chomba E, Patel A, Esamai F, Garces A, Althabe F, Kodkany B, Mabeya H, Manasyan A, Carlo WA, Derman RJ, Hibberd PL, Liechty EK, Krebs N, Hambidge KM, Buekens P, Moore J, Jobe AH, Koso-Thomas M, Wallace DD, Stalls S, Goldenberg RL; EMONC Trial Investigators. A combined community- and facility-based approach to improve pregnancy outcomes in low-resource settings: a Global Network cluster randomized trial. BMC Med. 2013 Oct 3;11:215. doi: 10.1186/1741-7015-11-215. PMID 24090370
- [Derived] Pasha O, Goldenberg RL, McClure EM, Saleem S, Goudar SS, Althabe F, Patel A, Esamai F, Garces A, Chomba E, Mazariegos M, Kodkany B, Belizan JM, Derman RJ, Hibberd PL, Carlo WA, Liechty EA, Hambidge KM, Buekens P, Wallace D, Howard-Grabman L, Stalls S, Koso-Thomas M, Jobe AH, Wright LL. Communities, birth attendants and health facilities: a continuum of emergency maternal and newborn care (the Global Network's EmONC trial). BMC Pregnancy Childbirth. 2010 Dec 14;10:82. doi: 10.1186/1471-2393-10-82. PMID 21156060
- See also: The Global Network for Women's and Children's Health Research website contains information regarding the EmONC Trial, as well as other Global Network studies. — http://gn.rti.org/